CLINICAL TRIAL: NCT04580264
Title: Lifestyle Online Re-Intervention On Eating Behaviour and BMI On Obese Hypertensive Patients
Brief Title: Online Re-Intervention On Eating Behaviour and BMI On Obese Hypertensive Patients
Acronym: LOREB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Juan F. Lisón Párraga, Dr, Professor of the Deparment of Biomedical Sciences, Cardenal Herrera University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNIVERSITY CARDENAL HERRERA-27
Record Dates: First submitted 2020-10-02; First posted 2020-10-08 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Hypertension; Overweight and Obesity
Keywords: Hypertension; Obesity; Internet; Re-intervention; Eating Behaviour; Physical Activity
MeSH Terms: conditions — Hypertension; Overweight; Obesity; Feeding Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): All participants will receive access to the same web-based lifestyle intervention (exercise and nutritional education)
  Interventions: Behavioral: REINTERVENTION

INTERVENTIONS:
Behavioral: REINTERVENTION — This self-applied online program will take three months and comprise 9 behavioural modules developed gradually, achieving the changes needed on eating and physical activity habits, supported by audiovisual instructions given by an hypertension specialist doctor.

SUMMARY:
This research will constitute a 3-year follow-up that includes a re-evaluation and re-intervention of overweight or obese adults suffering from hypertension, who already participated in a similar programme with the same objectives 3 years ago.

Patients will be recruited in the Hypertension Unit of a public hospital and assigned to a experimental group. The evaluation will include: eating behaviour, body mass index (BMI) and physical activity levels.

DETAILED DESCRIPTION:
Hypertension incidence and overweight or obesity related, constitute a worrying public health problem nowadays. Evidence indicates that, despite the existence of several factors involved in their etiology, diet and physical activity play a particularly important role in the treatment and prevention of obesity and associated disorders.

However, interventions for the treatment of obesity encounter some environmental and personal barriers, specifically problems or deficits in motivation. These barriers sometimes make it difficult to implement intervention strategies. In this sense, there is an important agreement about the need to generate alternatives and strategies which promote intrinsic motivation, self-regulation and self-efficacy as fundamental variables which have a direct relationship with the adherence and success of obesity treatments.

To achieve this, Information and Communication Technologies (ICTs) are a very promising alternative, as they can provide personalised feedback and can be flexibly adapted to each user. In addition, ICTs also present other important advantages, especially their excellent cost-benefit ratio, and the possibility of increasing the efficiency of the interventions, since they allow to reach a greater number of users at a lower cost.

This research will constitute a 3-year follow-up that includes a re-evaluation and re-intervention of overweight or obese adults suffering from hypertension, who already participated in a similar programme with the same objectives 3 years ago.

Patients will be recruited in the Hypertension Unit of a public hospital and assigned to a experimental group. The evaluation will include: eating behaviour, body mass index (BMI) and physical activity levels.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension.
* Overweight or obesity (25 ≤ BMI ≤ 35 kg/m2).
* Aged between 18-65 years.
* Being a participant of the program 3 years ago.

Exclusion Criteria:

* Not having access to the Internet or lack of information about it.
* Treatment with more than 3 antihypertensive drugs.
* Meet the criteria of the DSM-IV-TR of a Food Disorder.
* Presenting some type of severe psychiatric disorder.
* Disability that prevents or hinders physical exercise.
* Receiving some treatment for weight loss.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-19 (Actual)

PRIMARY OUTCOMES:
Eating Behaviour | 3 months
  Eating Behaviour will be measured with the DEBQ (Dutch Eating Behaviour Questionnaire). DEBQ evaluates eating behaviour that may contribute to or mitigate the development of overweight. It consists of 33 items, with a 5-point Likert scale, which 89 evaluate three eating styles. The Emotional Eating Scale has 13 items (e.g. "Do you have a desire to eat when you are angry?"), the External Eating Scale has 10 items (e.g. "Do you eat more than usual when you see others eating?"), and the Restrictive Eating Scale has 10 items (e.g. "Do you eat less deliberately so that you don't gain weight?").

SECONDARY OUTCOMES:
BMI | 3 Month
  Body Mass Index
Physical activity | 3 months
  Levels of physical activity (measured with Short-International Physical Activity questionnaire). This Questionnaire assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives are considered to estimate total physical activity in MET-min/week and time spent sitting.

CONTACTS AND LOCATIONS:
Overall Officials: JUAN FRANCISCO L PÁRRAGA, PhD, Principal Investigator — Cardenal Herrera University
Locations (1):
- Enrique Rodilla Sala, Sagunto, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lison JF, Palomar G, Mensorio MS, Banos RM, Cebolla-Marti A, Botella C, Benavent-Caballer V, Rodilla E. Impact of a Web-Based Exercise and Nutritional Education Intervention in Patients Who Are Obese With Hypertension: Randomized Wait-List Controlled Trial. J Med Internet Res. 2020 Apr 14;22(4):e14196. doi: 10.2196/14196. PMID 32286232